CLINICAL TRIAL: NCT02138006
Title: Stockholm Diabetes Intervention Study
Brief Title: Long-term Effects of Intensive Insulin Treatment in Type 1 Diabetes
Acronym: SDIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Nystrom, dr, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPN-2012
Record Dates: First submitted 2014-05-09; First posted 2014-05-14 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Heart Disease; Stroke; Renal Failure
MeSH Terms: conditions — Coronary Disease; Stroke; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive insulin treatment (Experimental): Intensive insulin treatment
  Interventions: Drug: Intensive insulin treatment
- Standard insulin treatment (Active Comparator): Standard insulin treatment
  Interventions: Drug: Standard insulin treatment

INTERVENTIONS:
Drug: Intensive insulin treatment — Mealtime insulin (Actrapid) Basal insulin (Monotard)
  Other Names: Basal-bolus insulin treatment
  Arms: Intensive insulin treatment
Drug: Standard insulin treatment — Insulin Mixtard
  Other Names: Mixed insulin 2-3 times per day
  Arms: Standard insulin treatment

SUMMARY:
To investigate long-term effects on cardiovascular mortality/morbidity and renal failure in type 1 diabetes patients former randomized to intensive insulin treatment

DETAILED DESCRIPTION:
The Stockholm Diabetes Intervention Study (SDIS) aimed to determine whether intensified insulin treatment were feasible and led to less serious diabetic complications. 102 patients with type 1 diabetes mellitus were randomized (October 1982 to March 1984) to intensified conventional treatment (ICT; n=48) or standard treatment (ST; n=54). The randomized SDIS study lasted for 7.5 years, whereas 96 patients were fully evaluated. Thereafter patients were assigned to their regular clinical visits.

In the present interventional study we wanted to study all-cause mortality and cardiovascular outcomes (i.e. myocardial infarction and stroke), and renal failure in the SDIS cohort until december 31 2011.

ELIGIBILITY:
Inclusion Criteria:

* Born 1930 or later
* Type 1 diabetes
* Nonproliferative retinopathy
* Normal serum creatinine
* Unsatisfactory blood glucose control

Exclusion Criteria:

* Alcohol/drug abuse
* Proliferative retinopathy

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 1982-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nyström, Md, PhD, Principal Investigator — Karolinska Institutet Dept of clinical science and education Södersjukhuset Stocholm
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Reichard P, Nilsson BY, Rosenqvist U. The effect of long-term intensified insulin treatment on the development of microvascular complications of diabetes mellitus. N Engl J Med. 1993 Jul 29;329(5):304-9. doi: 10.1056/NEJM199307293290502. PMID 8147960
- [Background] Jensen-Urstad KJ, Reichard PG, Rosfors JS, Lindblad LE, Jensen-Urstad MT. Early atherosclerosis is retarded by improved long-term blood glucose control in patients with IDDM. Diabetes. 1996 Sep;45(9):1253-8. doi: 10.2337/diab.45.9.1253. PMID 8772731
- [Background] Reichard P, Britz A, Cars I, Nilsson BY, Sobocinsky-Olsson B, Rosenqvist U. The Stockholm Diabetes Intervention Study (SDIS): 18 months' results. Acta Med Scand. 1988;224(2):115-22. doi: 10.1111/j.0954-6820.1988.tb16748.x. PMID 3048052
- [Background] Reichard P, Pihl M. Mortality and treatment side-effects during long-term intensified conventional insulin treatment in the Stockholm Diabetes Intervention Study. Diabetes. 1994 Feb;43(2):313-7. doi: 10.2337/diab.43.2.313. PMID 8288056
- [Background] Rathsman B, Jensen-Urstad K, Nystrom T. Intensified insulin treatment is associated with improvement in skin microcirculation and ischaemic foot ulcer in patients with type 1 diabetes mellitus: a long-term follow-up study. Diabetologia. 2014 Aug;57(8):1703-10. doi: 10.1007/s00125-014-3248-2. Epub 2014 May 7. PMID 24802206

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive Insulin Treatment | Standard Insulin Treatment
Started | 48 | 54
Completed | 48 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Insulin Treatment | Standard Insulin Treatment | Total
Number analyzed (Participants) | 48 | 54 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 54 | 102
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (8) | 32 (7) | 31 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 22 | 26 | 48
Region of Enrollment [Number; unit: participants]
  Sweden | 48 | 54 | 102

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Mortality
Description: All cause mortality and composite mortality from myocardial infarction, stroke and renal failure
Time Frame: Up to 28 years
Measure: Number; unit: participants
Arm/Group | Intensive Insulin Treatment | Standard Insulin Treatment
Number analyzed (Participants) | 48 | 54
participants | 7 | 11
Statistical Analysis 1: Comparison: Intensive Insulin Treatment vs Standard Insulin Treatment; Test type: Superiority or Other; p = 0.30, Log Rank

2. Secondary Outcome: Morbidity of Cardiovascular Complications
Description: Morbidity of: coronary heart disease, stroke and renal failure
Time Frame: Up to 28 years
Measure: Number; unit: participants
Arm/Group | Intensive Insulin Treatment | Standard Insulin Treatment
Number analyzed (Participants) | 48 | 54
participants | 6 | 11

ADVERSE EVENTS:
Arm/Group | Intensive Insulin Treatment | Standard Insulin Treatment
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/54
Other Adverse Events (participants affected / at risk) | 0/48 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes